ISN/Protocol 8951-CL-0301

# PATIENT REPORTED OUTCOME STATISTICAL ANALYSIS PLAN

Version 2.0

02-MAY-2023

A Phase 3, Global, Multi-Center, Double-Blind, Randomized, Efficacy Study of Zolbetuximab (IMAB362) Plus mFOLFOX6 Compared with Placebo Plus mFOLFOX6 as First-line Treatment of Subjects with Claudin (CLDN)18.2-Positive, HER2-Negative, Locally Advanced Unresectable or Metastatic Gastric or Gastroesophageal Junction (GEJ) Adenocarcinoma

Spotlight

ISN/Protocol 8951-CL-0301

Sponsor:
Astellas Pharma Global Development, Inc. (APGD)

1 Astellas Way
Northbrook, IL 60062

This document contains confidential information which is the intellectual property of Astellas. By accepting or reviewing this document, you agree to hold this information in confidence and not copy or disclose it to others or use it for unauthorized purposes except (1) as otherwise agreed to in writing; (2) where required by applicable law; (3) where disclosure is directly related to the care and safety of the research participant; and (4) where disclosure of such information is made to a member of the investigator's team who agrees to hold this information in confidence.

02-May-2023 Astellas Page 1 of 41

## **Table of Contents**

| 1 | INT | TRODUCTION | 5 |
|---|---|---|---|
| | 1.1 | Objectives of the COA Analysis · | 5 |
| | 1.2 | Study Objectives · | 6 |
| | 1.2.1 | Primary Objective · | 6 |
| | 1.2.2 | Secondary Objectives · | 6 |
| | 1.2.3 | Exploratory Objectives · | 6 |
| | 1.3 | Study Design···· | 6 |
| | 1.4 | COA Instruments····· | 8 |
| | 1.4.1 | EORTC QLQ-C30 ····· | 9 |
| | 1.4.2 | EORTC QLQ-OG25 ····· | 9 |
| | 1.4.3 | GP | 9 |
| | 1.4.4 | EQ-5D-5L ····· | 9 |
| | 1.4.5 | Assessment Schedule · | _ |
| 2 | AN. | ALYSIS SETS ····· | 10 |
| 3 | AN | ALYSIS VARIABLES ····· | 10 |
| | 3.1 | General Variables and Derivations | 10 |
| | 3.1.1 | Study Day · | 10 |
| | 3.1.2 | Baseline | |
| | 3.1.3 | Derived Timepoints · | |
| | 3.1.4 | Other Derivations · | |
| | 3.2 | PRO Variables · | 11 |
| | 3.2.1 | Variables generated from QLQ-C30 ····· | 11 |
| | 3.2.2 | Variables Generated From QLQ-OG25 ······ | 14 |
| | 3.2.3 | Variables Generated From GP ····· | 16 |
| | 3.2.4 | Variables Generated From EQ-5D-5L · | |
| | 3.3 | Time to PRO Deterioration · | 18 |
| | 3.3.1 | Time To First Clinically Meaningful Deterioration (TTFD) · | 18 |
| | 3.3.2 | Time To First Confirmed Clinically Meaningful Deterioration (TTFCD) · · · | 19 |
| | 3.3.3 | Time To Definitive Clinically Meaningful Deterioration (TTDD) · | 20 |
| | 3.3.4 | Summary Of Time to PRO Deterioration Analysis · | |
| | 3.4 | Subgroups of Interest · | 21 |
| 4 | STA | ATISTICAL ANALYSES ····· | 21 |
| | 4.1 | General Considerations | 21 |

| | 4.2 | Handling of Missing Data · · · · · · 21 |
|---|-------|---------------------------------------------------------------|
| | 4.2.1 | Missing Items ······21 |
| | 4.2.2 | Missing Forms · · · · · 21 |
| | 4.3 | Study Participants · · · · · · 22 |
| | 4.3.1 | Participant Disposition · · · · · · 22 |
| | 4.3.2 | PRO Completion · · · · · 22 |
| | 4.3.3 | Demographic and Other Baseline Characteristics · · · · · · 22 |
| | 4.4 | Descriptive Analyses · · · · · 23 |
| | 4.4.1 | Item Level · · · · · · 23 |
| | 4.4.2 | Domain and Overall Score Level · · · · · · 23 |
| | 4.5 | Longitudinal Analysis of Change From Baseline · · · · · · 23 |
| | 4.5.1 | Mixed Model Repeated Measures ······23 |
| | 4.6 | Responder Analysis · · · · · · 25 |
| | 4.7 | Time to Event Analysis · · · · · · 25 |
| | 4.7.1 | Sensitivity Analyses ·······26 |
| | 4.8 | Subgroup Analyses······27 |
| 5 | SUI | PPORTING DOCUMENTATION ······28 |
| | 5.1 | Appendix A List of Abbreviations ······28 |
| | 5.2 | Appendix B QLQ-C30·····29 |
| | 5.3 | Appendix C QLQ-OG25 ············33 |
| | 5.4 | Appendix D GP······36 |
| | 5.5 | Appendix E EQ-5D-5L · · · · · · · 37 |
| 6 | REI | FERENCES39 |
| 7 | SIG | NATURE ················41 |

## **PRO SAP Version History Summary**

The changes from the prior approved SAP that impact analyses are listed with the rationale in the table below.

| PRO<br>SAP<br>Version | Approval<br>Date | SAP<br>Section(s) | Change | Rationale |
|---|---|---|---|---|
| 1.0 | 09-MAR-2022 | | Not Applicable | Original Version |
| 2.0 | 02-MAY-<br>2023 | 1.4.1 | Added note on EORTC<br>QLQ-C30 recall period<br>Removed analysis visit<br>window section | 1.4.1 Correction 3.1.4 and 4.7 Alignment |
| | | 3.1.4 | | with the clinical SAP |
| | | 3.2.1 | EORTC QLQ-C30 threshold correction | 3.2.1 and 3.2.2 Update to the thresholds |
| | | 3.2.2 | EORTC QLQ-OG25<br>threshold correction | 3.2.4 Updated EQ-5D-5L utility index mapping |
| | | 3.2.4 | Updated EQ-5D-5L mapping function | function based on NICE recommendation |
| | | 4.5 | Updated MMRM | 4.5 and 4.6 Updated based |
| | | 4.6 Updated responder analyses | on sample size and predictions at Cycle 9 Day 1 | |
| | | 4.7 | Retained and specified one-sided test for the 3 key scores in time to | 6 Reference corrections Appendix F Removed based on section 3.2.4 edits |
| | | | event analyses | |
| | | 6 and pg 16,<br>18, and 19 | Minor corrections to references | |
| | | Appendix F | Deleted | |

ISN/Protocol 8951-CL-0301

#### 1 INTRODUCTION

This document describes the rules and conventions to be used in the presentation and analysis of clinical outcome assessment (COA) data for Protocol 8951-CL-0301. It describes the data to be summarized and analyzed, including specifics of the statistical analyses to be performed.

This statistical analysis plan (SAP) is based on protocol version 6.0 dated 29 Sep 2021 and amendment 5.

This plan may be revised during the study to accommodate protocol amendments and/or to make changes to adapt to unexpected issues in study execution and/or data that affect planned analyses. The final plan, if revised, will document all changes and be issued prior to database lock.

## 1.1 Objectives of the COA Analysis

The aim of this project is to perform in-depth statistical analyses on the patient-reported outcomes (PROs) data collected in the 8951-CL-0301 study. This is to address protocolspecific objective COA-related as specified in section 3.1.

The objective of the COA efficacy analysis is to enhance the understanding of the benefits of zolbetuximab when combined with mFOLFOX6 compared to placebo and mFOLFOX6 on disease-related symptoms, pain, and health related quality of life (HRQoL) in patients with Claudin (CLDN) 18.2-positive, HER2-negative, locally advanced unresectable or metastatic gastric or Gastroesophageal Junction (GEJ) adenocarcinoma. Treatment effects on symptoms, pain, HRQoL, function, and health status as measured by the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire EORTC QLQ-C30, EORTC Quality of Life Questionnaire - Oesophago-Gastric Module EORTC QLQ-OG25, Global Pain (GP), and the EuroQoL 5 dimension-5 level (EQ-5D-5L) instruments will be further evaluated by examining:

- Longitudinal change from baseline
- Time to first clinically meaningful deterioration (TTFD) in symptoms prior to disease progression
- Time to confirmed clinically meaningful deterioration (TTCD) in symptoms prior to disease progression
- Time to definitive clinically meaningful deterioration (TTDD) in symptoms prior to disease progression
- Proportion of patients with improvement/no change/deterioration in symptoms and HRQoL

Analysis will be performed for all scales of the above PRO instruments, except for certain analysis on physical functioning (PF) and Global Health Status (GHS)/Quality of Life (QoL) from EORTC QLQ-C30, and the EORTC QLQ-OG25 Pain which are analyzed in the clinical

SAP (Version 2.0, dated 18Nov2021). These exceptions will be specified in the corresponding sections.

### 1.2 Study Objectives

#### 1.2.1 Primary Objective

The primary objective is to evaluate the efficacy of zolbetuximab plus mFOLFOX6 compared with placebo plus mFOLFOX6 (as first-line treatment) as measured by progression free survival (PFS) in subjects with CLDN 18.2-positive, HER2-negative locally advanced unresectable or metastatic gastric and GEJ adenocarcinoma.

#### 1.2.2 Secondary Objectives

The secondary objectives are:

- To evaluate efficacy as measured by overall survival (OS) as a key secondary objective
- To evaluate the physical function (PF), OG25-Pain and GHS/QoL scores as measured by EORTC as a key secondary objective
- To evaluate efficacy as measured by objective response rate (ORR)
- To evaluate efficacy as measured by duration of response (DOR)
- To evaluate safety and tolerability of zolbetuximab
- To further evaluate other health related quality of life (HRQoL) using additional parameters as measured by EORTC QLQ-C30, QLQ-OG25, Global Pain (GP), and the EuroQoL 5 dimension-5 level (EQ-5D-5L) questionnaires
- To evaluate the pharmacokinetics of zolbetuximab
- To evaluate the immunogenicity profile of zolbetuximab.

#### 1.2.3 Exploratory Objectives

The exploratory objectives are:

- To evaluate efficacy as measured by time to progression (TTP)
- To evaluate PFS following subsequent anti-cancer treatment (PFS2)
- To evaluate disease control rate (DCR)
- To evaluate potential genomic and /or other biomarkers that may correlate with treatment outcome to zolbetuximab and mFOLFOX6
- To evaluate health resource utilization (HRU).

## 1.3 Study Design

This is a global, multi-center, double-blind, 1:1 randomized, phase 3 study evaluating the efficacy of zolbetuximab plus mFOLFOX6 versus placebo plus mFOLFOX6 as first-line

treatment in subjects with CLDN 18.2-positive, HER2-negative locally advanced unresectable or metastatic gastric and GEJ adenocarcinoma.

Approximately 550 subjects will be 1:1 randomized into 1 of 2 treatment arms:

- Arm A (mFOLFOX6 chemotherapy in combination with zolbetuximab)
- Arm B (mFOLFOX6 chemotherapy in combination with placebo).

The randomization will be stratified by:

- Region (Asia vs Non-Asia)
- Number of metastatic sites (0 to 2 vs  $\ge$ 3)
- Prior gastrectomy (Yes or No).

Subjects will be treated with either zolbetuximab (Arm A) or placebo (Arm B) on Days 1 and 22 starting at Cycle 1 Day 1 (C1D1) until the subject meets study treatment discontinuation criteria. Subjects will also receive 12 treatments of mFOLFOX6 (or components of mFOLFOX6 if some components are discontinued due to toxicity) over 4 cycles (1 cycle = 42 days) on Days 1, 15, and 29 of each cycle. After 12 mFOLFOX6 treatments, subjects may continue to receive 5-FU (fluorouracil) and folinic acid on Days 1, 15 and 29 of each cycle at the investigator's discretion until the subject meets study treatment discontinuation criteria.

If a subject discontinues mFOLFOX6 (or its components) due to any reason other than disease progression as confirmed by independent review committee (IRC), they may continue on zolbetuximab/placebo and continue to follow the study treatment period schedule of assessments at the discretion of the investigator provided that the following have been met:

- the subject completed at least 1 cycle (42 days) of mFOLFOX6 treatment;
- the subject will not receive anoother systemic chemotherapy, immunotherapy, radiotherapy or other treatment intended for antitumor activity; and
- in the investigator's opinion the subject continues to derive clinical benefit with acceptable toxicity.

Following discontinuation from zolbetuximab/placebo, subjects will have a study treatment discontinuation visit, and 30-day and 90-day safety follow-up visits following their last dose of zolbetuximab/placebo. Additionally, if mFOLFOX6 (all components) is discontinued on a different day than zolbetuximab/placebo, subjects will also have a study treatment discontinuation visit, and 30-day and 90-day safety follow-up visits following the last dose of mFOLFOX6.

If a subject discontinues all study treatments (zolbetuximab/placebo and all components of mFOLFOX6) prior to disease progression, the subject will enter the post-treatment follow-up period and continue to undergo scheduled imaging assessments every 9 weeks until radiologic disease progression or until the subject starts any other anti-cancer treatment, whichever occurs earlier.

If study treatment (zolbetuximab/placebo and all components of mFOLFOX6) is discontinued due to disease progression, the subject will enter the long-term and survival follow-up period. Survival follow-up period will continue until death from any cause.

HRQoL and HRU will be assessed during the visit (or up to 48 hours) before any antiemetic or drug treatment(s) administration and before the disease status is discussed with the subject. Assessments will be collected at Screening (except HRU), every 3 weeks, at study treatment discontinuation and 30 and 90 days post-zolbetuximab/placebo treatment.

The study schema is provided in Figure 1.

Figure 1 Study Schema



Notes: 5-FU: fluorouracil; CLDN: Claudin; HER2: human epidermal growth factor receptor 2; IRC: independent review committee; mFOLFOX6: 5-fluorouracil, folinic acid and oxaliplatin; RECIST: Response Evaluation Criteria in Solid Tumors.

#### 1.4 COA Instruments

Patient-reported outcomes will be assessed through four different instruments:

- European Organization for Research and Treatment of Cancer Quality of Life Core 30: EORTC QLQ-C30
- EORTC Quality of Life Questionnaire Oesophago-Gastric Module: EORTC QLQ-OG25
- Global Pain (GP)
- EuroQoL 5 dimension-5 level (EQ-5D-5L).

#### 1.4.1 **EORTC QLQ-C30**

The EORTC QLQ-C30 instrument (Aaronson et al, 1993) is a generic questionnaire consisting of 30 items developed to assess symptoms and functioning of cancer patients. The instrument yields 5 functional scales, 4 symptom scales, 1 global health status (GHS) / quality of life (QoL) scale and 1 financial impact score. Most items are scored 1 ("not at all") to 4 ("very much") except for the items contributing to the global health status/QoL, which are scored 1 ("very poor") to 7 ("excellent"). The recall period for each question is "during the past week" (note a recall period is not indicated for questions 1-5). An outcome variable consisting of a score from 0 to 100 is derived for each of the scales. Higher scores on symptoms indicate a worse health state. Higher scores on the global health status and functioning scales indicate better health status/function.

The QLQ-C30 is presented in Appendix B QLQ-C30.

#### 1.4.2 EORTC QLQ-OG25

The QLQ-OG25 is a 25-item instrument that evaluates gastric and GEJ cancer-specific symptoms such as stomach discomfort, difficulties eating and swallowing, and indigestion. This module consists of 6 scales: dysphagia, eating restrictions, reflux, odynophagia, pain and discomfort, and anxiety, as well as 10 single items. Each item is rated on a four-point Likert scale ranging from 1 = "not at all" to 4 = "very much".

The QLQ-OG25 is presented in Appendix C QLQ-OG25.

#### 1.4.3 GP

The GP is a single assessment of overall pain on a scale from 0 (no pain) to 10 (pain as bad as you can imagine).

The GP is presented in Appendix D GP.

#### 1.4.4 EQ-5D-5L

The EQ-5D-5L is a quality of life (QoL) instrument for self-reported assessment of 5 domains of health: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each domain is rated by selecting 1 of 5 standardized categorizations ranging from 'no problem' to 'extreme problem'. The final question is a visual analogue scale (VAS) to rank health status from best health imaginable (100) to worst health imaginable (0).

The EQ-5D-5L is presented in Appendix E EQ-5D-5L and Appendix F Utility Index calculation (EQ-5D-5L).

#### 1.4.5 Assessment Schedule

The assessment schedule for the PRO instruments is provided in Table 1.

ISN/Protocol 8951-CL-0301

**Table 1 PRO Instruments Assessment Schedule** 

| | | Stud | Study Treatment Period (Each Cycle = 42 days) | | | | | ays) | ] | Follow- | up Per | riod <sup>b</sup> | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Study Day | Screening | Cycles 1 to 4 Zolbetuximab/Placebo + mFOLFOX6 | | | Cycle 5+ Zolbetuximab/Placebo + 5FU+Folinic Acid | | Study<br>Discontinuation | 30-Day Follow-up<br>Visit | 90-Day Follow-up<br>Visit | Post Treatment<br>Follow-up | Long Term and<br>Survival Follow-up <sup>b</sup> | | | |
| | | 1 | 15 | 22 | 29 | 1 | 15 | 22 | 29 | | | | | |
| Window<br>(Days) | -45 to -1 | 0 | +5 | +5 | +5 | +5 | +5 | +5 | +5 | +7 | +7 | +7 | ±7 | ±14 |
| PRO<br>Assessments <sup>a</sup> | X | X | | X | | X | | X | | X | X | X | | |

<sup>&</sup>lt;sup>a</sup> PRO instruments are to be administered on IMAB362/placebo visit days before any antiemetic or drug treatment or other scheduled assessments are conducted and before the disease status is discussed with the subject.

#### 2 ANALYSIS SETS

All PRO analyses described in this SAP will be performed on the Full Analysis Set (FAS) as defined in the clinical SAP (Version 2.0, dated 18Nov2021), i.e. all subjects who are randomized to 1 of the treatment arms. All subjects will be analyzed as randomized (not by actual treatment received). FAS in this study is identical to intent-to-treat (ITT) set.

#### 3 ANALYSIS VARIABLES

#### 3.1 General Variables and Derivations

#### 3.1.1 Study Day

Study day as defined in the clinical SAP (Version 2.0, dated 18Nov2021) will be used. The study day will be calculated in reference to the date of the first dose of study drug. Treatment Day 1 corresponds to the date the subject received the first dose of study drug. For assessments conducted on or after the date of the first dose of study drug, study day will be calculated as (assessment date - date of first dose of study drug) + 1.

#### 3.1.2 Baseline

The baseline measurement is the last measurement taken prior to initial study drug administration (i.e., Cycle 1 Day 1 pre-dose assessment). Both date and time of drug administration and measurement should be considered to identify the baseline value. If the

<sup>&</sup>lt;sup>b</sup> If a subject discontinues all study treatments (IMAB362/placebo and all components of mFOLFOX6) prior to IRC confirmed disease progression, the subject will enter the post-treatment follow-up period and continue to undergo imaging assessment every 9 weeks (or every 12 weeks if subjects has been on study over 54 weeks) until radiologic disease progression (i.e., PFS) or the subject starts subsequent anti-cancer treatment, whichever occurs earlier. If study treatment (IMAB362/placebo and all components of mFOLFOX6) is discontinued due to PD, the subject will enter the Long term and survival follow-up period.

time is not available, then only the date will be used, and it will be assumed that assessments on day 1 were administered prior to dosing.

The post-baseline value is defined as a measurement taken after initial study drug administration.

Change from baseline is defined as (post baseline value - baseline value).

#### 3.1.3 Derived Timepoints

All timepoints will be used as in the ADaM datasets received by the sponsor.

#### 3.1.4 Other Derivations

No other derivations besides PRO endpoints will be described in this analysis plan.

#### 3.2 PRO Variables

#### 3.2.1 Variables generated from QLQ-C30

The EORTC QLQ-C30 scale scores will be calculated using the EORTC QLQ-C30 Scoring Manual (Fayers et al, 2001). The instrument yields the following scales: Global health status/Quality of Life (QL2; 2 items; score range 0-100).

- Functional scales:
  - o Physical functioning (PF2; 5 items; score range 0-100)
  - o Role functioning (RF2; 2 items; score range 0-100)
  - o Emotional functioning (EF; 4 items; score range 0-100)
  - o Cognitive functioning (CF; 2 items; score range 0-100)
  - o Social functioning (SF; 2 items; score range 0-100)
- Symptom scales/items:
  - o Fatigue (3 items; score range 0-100)
  - Nausea and vomiting (2 items; score range 0-100)
  - o Pain (2 items; score range 0-100)
  - O Dyspnea (1 item; score range 0-100)
  - o Insomnia (1 item; score range 0-100)
  - o Appetite loss (1 item; score range 0-100)
  - o Constipation (1 item; score range 0-100)
  - o Diarrhea (1 item; score range 0-100)
- Financial difficulties (1 item; score range 0-100)

ISN/Protocol 8951-CL-0301

Although not included in the original scoring manual (Fayers et al, 2001), it has been suggested in the literature that a single summary score can also be calculated for this instrument (Giesinger et al, 2016):

• Physical Functioning + Role Functioning + Social Functioning + Emotional Functioning + Cognitive Functioning + (100-Fatigue) + (100-Pain) + 100-(Nausea and Vomiting) + (100-Dyspnoea) + (100-Sleeping Disturbances) + (100-Appetite Loss) + (100-Constipation) + (100-Diarrhoea))/13.

The QLQ-C30 domain and single-item scores will be calculated according to the EORTC scoring manual presented in Appendix B QLQ-C30. The principle for scoring is the same for all scales. Briefly, outcome scores are computed by standardizing the average of the items (i.e., a raw score) making up the scale. Outcome scores are computed using a linear transformation of the raw score such that scores range from 0 to 100. A higher score represents a higher ("better") level of functioning, or a higher ("worse") level of symptoms, i.e., a high score for a functional scale represents a high/healthy level of functioning, a high score for the GHS represents a high QoL, but a high score for a symptom scale/item represents a high level of symptomatology/problems. Note that the global health status scale is based on only the 2 specific HRQoL items and not the entire questionnaire.

If at least half the items of a scale are present for a timepoint then the score will be calculated using the average of all items answered; otherwise the score will be set to missing. For single measures, if the item is missing the scale score is set to missing.

Physical and role functioning, as well as the global QoL revised scales are those that have been changed since version 1.0, and their short names are indicated a suffix "2" – for example, PF2, according to the instrument's manual (Fayers et al, 2001).

All the below definitions apply to all domains, except for the FI that will not be analyzed.

Change from baseline defined as post-baseline value minus baseline value will be calculated for each assessment for each scale and item.

Post-baseline item scores will be classified as according to the following item response categories:

- Worsening 3 points compared to baseline
- Worsening 2 points compared to baseline
- Worsening 1 point compared to baseline
- Stable
- Improved 1 point compared to baseline
- Improved 2 points compared to baseline
- Improved 3 points compared to baseline

**Sponsor: Astellas** ISN/Protocol 8951-CL-0301

Change in symptoms/functioning/global health status from baseline will be categorized as improvement/stable/deterioration using threshold values for change scores that connote clinically meaningful changes for patients.

Two sets of values will be used. For QL2 and PF, the primary threshold for deterioration will be derived by anchor-based analysis of the trial's data before data base lock occurs, as described in the 8951-CL-0303 study analysis plan (Version 1.0, dated 09Mar2022). For the rest of the domains, the primary threshold values will be based on values developed by Cocks et al. 2012 and shown in Table 3.

Table 2 Primary responder definition for EORTC QLQ-C30

| Score | Deterioration | Stable | Improvement |
|--------------------------|---------------|------------|-------------|
| Global health status/QoL | < -10 | -10 to +8 | >+8 |
| Financial difficulties* | >+10 | -10 to +3 | <-3 |
| <b>Functional scales</b> | | | |
| Physical functioning | < -10 | -10 to +7 | >+7 |
| Role functioning | <-14 | -14 to +12 | >+12 |
| Cognitive functioning | <-7 | -7 to +7 | >+7 |
| Emotional functioning | <-12 | -12 to +9 | >+9 |
| Social functioning | <-11 | -11 to +8 | >+8 |
| Symptom scales | | | |
| Fatigue | >+10 | +10 to -9 | <-9 |
| Pain | >+11 | +11 to -9 | <-9 |
| Nausea and vomiting | >+11 | +11 to -9 | <-9 |
| Diarrhea | >+15 | +15 to -11 | <-11 |
| Constipation | >+15 | +15 to -10 | <-10 |
| Appetite loss | >+14 | +14 to -13 | <-13 |
| Dyspnea | >+11 | +11 to -9 | <-9 |
| Insomnia | >+9 | +9 to -9 | <-9 |

<sup>\*</sup>FI will not be analyzed in this analysis plan.

For the sensitivity threshold as there were no other threshold values connoting clinically meaningful within-patient change identified in the literature, it will be based on the next highest value that will provide a different classification for deterioration and improvement to the primary one. The reason of this approach is that EORTC values are discrete in nature due to the transformation of raw scores to 0-100, therefore not all values are possible and certain threshold values will result in the same categorization for patients, e.g., for a single-item domain such as appetite loss, the possible values are 0, 33.3, 66.7 and 100, therefore a applying a threshold of 15 and 30 will result in the same classification of patients into responder categories. The sensitivity values for all domains are shown in Table 4.

**Sponsor: Astellas** ISN/Protocol 8951-CL-0301

Table 3 Sensitivity responder Definition for EORTC QLQ-C30

| Score | Deterioration | Stable | Improvement |
|--------------------------|---------------|------------|-------------|
| Global health status/QoL | <-17 | -17 to +8 | >+9 |
| Financial difficulties* | >+34 | -34 to +34 | <-34 |
| Functional scales | | | |
| Physical functioning | < -14 | -14 to +14 | >+14 |
| Role functioning | <-17 | -17 to +17 | >+17 |
| Cognitive functioning | <-17 | -17 to +17 | >+17 |
| Emotional functioning | <-17 | -17 to +17 | >+17 |
| Social functioning | <-17 | -17 to +17 | >+17 |
| Symptom scales | | | |
| Fatigue | >+12 | +12 to -12 | <-12 |
| Pain | >+17 | +17 to -17 | <-17 |
| Nausea and vomiting | >+17 | +17 to -17 | <-17 |
| Diarrhea | >+34 | +34 to -34 | <-34 |
| Constipation | >+34 | +34 to -34 | <-34 |
| Appetite loss | >+34 | +34 to -34 | <-34 |
| Dyspnea | >+34 | +34 to -34 | <-34 |
| Insomnia | >+34 | +34 to -34 | <-34 |

## 3.2.2 Variables Generated From QLQ-OG25

There will be six domains and ten single-item scores calculated for QLQ-OG25:

- Domain Scale Scores
  - o Dysphagia (3 items; score range 0-100)
  - o Eating restrictions (4 items; score range 0-100)
  - o Reflux (2 items; score range 0-100)
  - Odynophagia (2 items; score range 0-100)
  - o Pain and discomfort (2 items; score range 0-100)
  - o Anxiety (2 items; score range 0-100)
- Single Items Scores
  - o Eating in front of others (1 item; score range 0-100)
  - o Dry mouth (1 item; score range 0-100)
  - o Trouble with taste (1 item; score range 0-100)
  - o Body image (1 item; score range 0-100)
  - o Trouble swallowing saliva (1 item; score range 0-100)
  - Choked when swallowing (1 item; score range 0-100)

ISN/Protocol 8951-CL-0301

- o Trouble with coughing (1 item; score range 0-100)
- o Trouble talking (1 item; score range 0-100)
- Weight loss (1 item; score range 0-100)
- Hair loss (1 item; score range 0-100)

The QLQ-OG25 domain and single-item scores will be calculated according to the EORTC scoring manual presented in Appendix C QLQ-OG25. Raw scores will be transformed into a linear scale ranging from 0 to 100, with a high score for representing a higher ("worse") level of symptomatology/problems.

Change from baseline defined as post-baseline value minus baseline value will be calculated for each assessment for each scale and item.

Post-baseline item scores will be classified as according to the same item response categories described in section 3.1.2.

Post-baseline multi-item and single-item scale scores will be classified as improvement/no change/deterioration according to baseline scores at each assessment using a threshold to connote important change to subjects as follows:

- Improvement: a change from baseline ≤ -threshold points;
- Deterioration: a change from baseline ≥ threshold points
- No change: a change from baseline between (–threshold to threshold).

Literature reporting clinically important thresholds were not found. Two sets of values will be used. The primary threshold values will be obtained using the baseline distributions of QLQ-OG25 scores (e.g., a change equal to or greater than one-half the baseline standard deviation (SD) pooled over the two treatment arms) (Norman et al 2003, Sloan et al 2005) or a 1-category change in 1 item in the scale, whichever is larger. Sensitivity analysis will be performed using the next higher threshold that results in a different classification of patients into improvement, stable and deterioration categories as compared to the primary threshold, as for EORTC QLQ-C30.

The thresholds to be used for QLQ-OG25 scores are presented in Table 5. Number in parenthesis for primary threshold represents how change in 1 item corresponds to the 0-100 score of the scale.

Table 4 Predefined threshold values for QLQ-OG25

| QLQ-OG25 outcome | Primary threshold | Sensitivity threshold |
|---|---|---|
| • Dysphagia (3 items) | • 4-item scale: max (pooled | Next higher threshold that results in a |
| • Eating restrictions (4 items) | baseline ½ SD, 8.3) | different classification as compared to |
| • Reflux (2 items) | • 3-item scale: max (pooled | the primary threshold |
| • Odynophagia (2 items) | baseline ½ SD, 11.1) | |
| • Pain and discomfort (2 items) | • 2-item scale: max (pooled | |
| • Anxiety (2 items) | baseline ½ SD, 16.7) | |
| • Eating in front of others (1 | • 1-item scale: max (pooled | |
| item) | baseline ½ SD, 33.3) | |

ISN/Protocol 8951-CL-0301

| QLQ-OG25 outcome | Primary threshold | Sensitivity threshold |
|--------------------------------|-------------------|-----------------------|
| • Dry mouth (1 item) | | |
| • Trouble with taste (1 item) | | |
| • Body image (1 item) | | |
| • Trouble swallowing saliva (1 | | |
| item) | | |
| • Choked when swallowing (1 | | |
| item) | | |
| • Trouble with coughing (1 | | |
| item) | | |
| • Trouble talking (1 item) | | |
| • Weight loss (1 item) | | |
| • Hair loss (1 item) | | |

#### 3.2.3 Variables Generated From GP

The GP is a single assessment of overall pain on a scale ranging from 0 (no pain) to 10 (pain as bad as you can imagine). The score will be the numeric endorsement on the scale.

A higher score indicates a higher degree of pain.

Pain severity at baseline is defined as described in Table 6.

Table 5 Pain severity at baseline definition

| Severity level | Definition |
|---|---|
| Asymptomatic subjects | Subjects with a score of 0 at the baseline visit |
| Mildly symptomatic subjects | Subjects with a score of 1 to 4 at the baseline visit |
| Moderate symptomatic subjects | Subjects with a score of 5 or 6 at the baseline visit |
| Severely symptomatic subjects | Subjects with a score of 7 to 10 at the baseline visit |

Change from baseline defined as post-baseline value minus baseline value will be calculated for each assessment for each scale and item.

Post-baseline GP score will be classified as improvement/no change/deterioration according to baseline scores at each assessment using a threshold to connote important change to subjects as follows:

- Improvement: a change from baseline ≤ -threshold points;
- Deterioration: a change from baseline ≥ threshold points
- No change: a change from baseline between (–threshold to threshold).

Cut-off values of 2-point or greater change on a 11-point numerical pain rating scale have been proposed in the literature to detect clinically important changes in adults (Farrar, et al. 2000, Kendrick, et al. 2005). However, the use of these values in defining pain progression on the GP in subjects with CLDN18.2-positive, HER2-negative locally advanced unresectable or metastatic gastric and GEJ adenocarcinoma has not yet been validated. Therefore, a sensitivity analysis will be performed using a threshold obtained using the

ISN/Protocol 8951-CL-0301

baseline distributions of GP score (e.g., a change equal to or greater than one-half the baseline SD pooled over the two treatment arms) (Norman et al 2003; Sloan et al 2005).

The thresholds to be used for GP scores are presented in Table 7.

Table 6 Predefined thresholds for GP

| GP outcome | Primary threshold | Sensitivity threshold |
|------------|-------------------|-----------------------|
| Pain item | 2 points | Pooled baseline ½ SD |

#### 3.2.4 Variables Generated From EQ-5D-5L

A unique EQ-5D-5L health state is defined by combining 1 level from each of the 5 dimensions: this defines a profile that is primarily reported as a 5-digit number, for instance 11221. A total of 3125 possible health states are defined in this way. For example, state 11111 indicates no problems on any of the 5 dimensions, while state 12345 indicates no problems with mobility, slight problems with washing or dressing, moderate problems with doing usual activities, severe pain or discomfort and extreme anxiety or depression.

The instrument was specifically designed to provide an overall single number, called a weighted index, for each of the health states resulting from the combination of item responses (Dolan 1997). The weighted index constitutes a measure of utility, an economics term used to describe consumer preferences or in the present case patient preferences for different HRQoL states. The weighted index can be only derived from patients who have provided a complete 5-response profile. A higher index indicates better QoL.

The mapping (crosswalk) function developed by Hernández Alava et al (2017) will be used as UK's National Institute of Health and Care Excellence in a position statement (NICE 2019) does not recommend to use the EQ-5D-5L value set for England published by Devlin et al (2017) to derive utility values for their evidence submissions and according to the latest NICE health technology evaluations manual (NICE 2022): "The mapping function developed by the Decision Support Unit (Hernández Alava et al 2017), using the 'EEPRU dataset' (Hernández Alava et al, 2020), should be used for reference-case analyses."

A higher score for the domains indicates worse QoL. In contrast, a higher score for EQ-5D VAS indicates better QoL.

Change from baseline defined as post-baseline value minus baseline value will be calculated for each assessment for the EQ-5D-5L VAS and utility index scores as well as for the individual domain items.

Post-baseline individual domain scores will be classified as according to the following item response categories:

- Worsening  $\geq$  3 points compared to baseline
- Worsening 2 points compared to baseline
- Worsening 1 point compared to baseline

ISN/Protocol 8951-CL-0301

- Stable
- Improved 1 point compared to baseline
- Improved 2 points compared to baseline
- Improved  $\geq$  3 points compared to baseline.

Post-baseline scores for EQ-5D-5L VAS and utility index will be classified as improvement/no change/deterioration according to baseline scores at each assessment using thresholds denoting clinically meaningful change to subjects as follows:

- Improvement: a change from baseline ≥ threshold points;
- Deterioration: a change from baseline ≤ threshold points
- No change: a change from baseline between (–threshold to +threshold).

Pickard et al (2007) reported a clinically meaningful change range of 7 to 10 for EQ-5D VAS score. The value 7 will be used in the primary analysis and the value of 10 will be used in a sensitivity analysis.

To be noted that no thresholds denoting clinically meaningful change to subjects have been reported in the literature for EQ-5D-5L utility index. Therefore, for each utility index score, a change threshold will be used based on the baseline distributions of EQ-5D-5L utility index score: a change equal to or greater than one-half the baseline SD (pooled over the two treatment arms) will be considered clinically meaningful, a definition that is well supported and accepted by the existing literature as a difference that is robust and likely significant to subjects (Norman et al, 2003; Sloan et al, 2005).

#### 3.3 Time to PRO Deterioration

Time to clinically meaningful symptom worsening or HRQoL deterioration (PRO deterioration) will be analysed for each domain separately as appropriate and as described in section 4.7. For convenience, a generic term "time to first clinically meaningful deterioration" (TTFD) will be used both for symptom worsening and HRQoL deterioration, with an understanding of a specific meaning depending on the domain analysed. Three definitions of TTD will be explored: time to first clinically meaningful deterioration (TTFD), time to first confirmed clinically meaningful deterioration (TTFCD), and time to definitive clinically meaningful deterioration (TTDD).

#### 3.3.1 Time To First Clinically Meaningful Deterioration (TTFD)

TTFD will be defined as the duration of time from the date of randomization to the date of the first deterioration in PRO scores of at least one threshold unit as compared to the baseline score.

For those subjects who experienced a first clinically meaningful deterioration, TTFD will be computed as follows and then converted to months:

TTFD = Date of assessment when first clinically meaningful deterioration of at least one threshold unit was observed – Date of randomization + 1

ISN/Protocol 8951-CL-0301

Patients who did not experience clinically meaningful deterioration prior to the end of follow-up, radiographic progression, or death (if not progressed before death) will be censored at the date of the last available PRO assessment (i.e., date of the last non-missing value). Patients with no baseline assessment, patients with no post-baseline assessments, or patients whose baseline scores do not allow for further deterioration will be censored at the date of randomization. Death or progression will not be considered deterioration events.

In addition, the above definition will be repeated where death (due to any cause) will be counted as a TTFD event if the subject does not experience PRO deterioration prior to death and where death occurs within 2 scheduled assessments (e.g., 42 days) after the last available PRO assessment; progression will not be considered deterioration event. Analyses will be also repeated by using the sensitivity clinically meaningful threshold as defined in section 3.2.

#### 3.3.2 Time To First Confirmed Clinically Meaningful Deterioration (TTFCD)

Time to first confirmed clinically meaningful deterioration (TTFCD) will be defined as the duration of time from the date of randomization to the date of the first clinically meaningful deterioration in PRO scores of at least one threshold unit as compared to the baseline score which is

- confirmed at the next consecutive scheduled visit or
- followed by drop out, resulting in monotone missing data.

For those patients who experienced a first confirmed clinically meaningful deterioration, TTFCD will be computed as follows and then converted to months:

TTFCD = Date of assessment when first confirmed clinically meaningful deterioration was observed – Date of randomization + 1

Patients who did not experience a confirmed clinically meaningful deterioration prior to the end of follow-up, radiographic progression, or death (if not progressed before death) will be censored at the date of the last available PRO assessment (i.e., date of the last non-missing value). Patients with no baseline assessment, patients with no post-baseline assessments, or patients whose baseline scores do not allow for further deterioration will be censored at the date of randomization. Death or progression will not be considered deterioration events.

In addition, the above definition will be repeated where death (due to any cause) will be counted as a TTFCD event if the subject does not experience PRO deterioration prior to death and where death occurs within 2 scheduled assessments (e.g., 42 days) after the last available PRO assessment; progression will not be considered deterioration event.

Analyses will be also repeated by using the sensitivity clinically meaningful threshold as defined in section 3.2.

ISN/Protocol 8951-CL-0301

### 3.3.3 Time To Definitive Clinically Meaningful Deterioration (TTDD)

TTDD will be defined as the duration of time from the date of randomization to the date of the first deterioration in PRO scores of at least one threshold unit as compared to the baseline score if the deterioration of at least one threshold unit as compared to the baseline score is:

- also observed at all time points thereafter (e.g., after the first deterioration is observed) or
- the patient dropped out after deterioration, resulting in missing data.

For those patients who experienced a definitive meaningful deterioration, TTDD will be computed as follows and then converted to months:

TTDD = Date of assessment when definitive clinically meaningful deterioration was observed – Date of randomization + 1

Patients who did not experience definitive clinically meaningful deterioration prior to the end of follow-up, radiographic progression, or death (if not progressed before death) will be censored at the date of the last available PRO assessment (i.e., date of the last non-missing value). Patients with no baseline assessment, patients with no post-baseline assessments, or patients whose baseline scores do not allow for further deterioration will be censored at the date of randomization. Death or progression will not be considered deterioration events.

In addition, the TTTD definition will be repeated where death (due to any cause) will be counted as an event if the subject does not experience PRO deterioration prior to death and where death occurs within 2 scheduled assessments (e.g., 42 days) after the last available PRO assessment; progression will not be considered deterioration event.

Analyses will be also repeated by using the sensitivity clinically meaningful threshold as defined in section 3.2 above.

#### 3.3.4 Summary Of Time to PRO Deterioration Analysis

A summary of all the definitions that will be explored is provided in the following table:

Table 7 Summary of time to PRO deterioration analysis

| <b>Definition</b> # | Description | Threshold | Death |
|---------------------|--------------------------|-------------|-----------|
| 1 | First deterioration | Primary | Excluding |
| 2 | First deterioration | Primary | Including |
| 3 | First deterioration | Sensitivity | Excluding |
| 4 | First deterioration | Sensitivity | Including |
| 5 | Confirmed deterioration | Primary | Excluding |
| 6 | Confirmed deterioration | Primary | Including |
| 7 | Confirmed deterioration | Sensitivity | Excluding |
| 8 | Confirmed deterioration | Sensitivity | Including |
| 9 | Definitive deterioration | Primary | Excluding |
| 10 | Definitive deterioration | Primary | Including |
| 11 | Definitive deterioration | Sensitivity | Excluding |
| 12 | Definitive deterioration | Sensitivity | Including |

ISN/Protocol 8951-CL-0301

### 3.4 Subgroups of Interest

The following subgroups may be considered:

- 1. Age category 1 (65 years or younger vs older than 65 years)
- 2. Region (Asia vs Non-Asia)

#### 4 STATISTICAL ANALYSES

#### 4.1 General Considerations

Continuous data will be described by the number of observations (N), the number of missing observations (Nmiss), mean, SD, median, first quartile (Q1), third quartile (Q3), minimum (min), maximum (max). Categorical data will be described by the number (n) and percentage (%) of patients in each category. Missing and invalid observations will be tabulated as separate categories. The calculation of proportions will not include the missing/invalid category.

For continuous data, the mean, median, Q1 and Q3 will be rounded to 1 additional decimal place compared to the original data. The SD will be rounded to 2 additional decimal places compared to the original data. Minimum and maximum will be displayed with the same accuracy as the original data.

For categorical data, percentages will be rounded to 2 decimal places.

For the PRO analyses, all summaries will be presented by treatment group, unless specified otherwise. Statistical comparisons will be made using two-sided tests at the  $\alpha$ =0.05 significance level unless stated otherwise. Due to the exploratory nature of the PRO analyses, adjustments for multiple comparisons will not be made.

Unless otherwise specified, all summaries will be presented by treatment group.

All data processing, summarization, and analyses will be performed using SAS Version 9.4 or higher (SAS Institute, North Carolina).

## 4.2 Handling of Missing Data

#### 4.2.1 Missing Items

In case of missing items, the domain and total scores will be calculated as indicated in the scoring manuals for each of the PRO instruments.

#### 4.2.2 Missing Forms

It is anticipated that the great majority of missing data in this study will have a monotone pattern, meaning that once a patient has missing data at one visit, data will be missing at all subsequent visits. There may be some small amount of intermittent (non-monotone) missing data (when patient skips intermediate visits but return for evaluations at subsequent visits).

ISN/Protocol 8951-CL-0301

The number and percentage of patients for each of the missing data patterns (no missing data, monotone missing data, and intermittent missing data) will be presented by treatment group.

Tabular summaries for the percentage of patients by the reason for discontinuation of study treatment, as well as for withdrawal from the study, will be provided in the clinical study report and will not be repeated herein. A plot of the mean score for the PRO scores over time by selected categories of discontinuation (including completers) will be provided. The reasons of discontinuation will be grouped as follows:

- Death
- Adverse event
- Disease relapse, lack of efficacy, and progressive disease
- Other.

## 4.3 Study Participants

#### 4.3.1 Participant Disposition

The subject disposition by treatment group for all PRO assessment time-points (e.g., analysis visits) will be provided:

- The number of subjects with PRO assessment expected
- The number and % of subjects with PRO assessment not expected due to progression
- The number and % of subjects with PRO assessment not expected due to death
- The number and % of subjects with PRO assessment not expected due to other reasons.

A PRO assessment is expected as long as the subject is alive and on treatment.

The subject disposition by treatment group per analysis visit will also be provided graphically by means of a stacked bar chart.

#### 4.3.2 PRO Completion

The PRO completion (unadjusted, i.e. over the FAS population) and compliance rates (adjusted, i.e. among expected patients at each assessment) will be presented in the clinical study report and will not be repeated here.

#### 4.3.3 Demographic and Other Baseline Characteristics

An extensive list of demographics and baseline disease characteristics is presented in the clinical SAP (Version 2.0, dated 18Nov2021), therefore these will not be repeated here.

ISN/Protocol 8951-CL-0301

### 4.4 Descriptive Analyses

#### 4.4.1 Item Level

For all items from all four instruments (QLQ-C30, QLQ-OG25, GP and EQ-5D-5L), the following will be provided:

- A table with the distribution of responses by treatment group at each assessment;
- A stacked column chart of the distribution of responses by treatment group at each assessment;
- A table with the distribution of change in response categories from baseline to each assessment by treatment group;
- A stacked column chart of the distribution of change in response categories from baseline to each assessment by treatment group.

#### 4.4.2 Domain and Overall Score Level

Domain and total scores will be summarized for the PRO instruments in the clinical study report and will not be repeated here.

A cumulative distribution plot showing a continuous plot of the absolute change from baseline during the study for the PRO scores on the X-axis and the cumulative percent of subjects experiencing that change on the Y-axis will be presented for the first six post-baseline visits. The presentation will be restricted to the first 6 post-baseline assessments and the following scales:

• EORTC QLQ-C30: GHS/QoL and PF and OG25-Pain.

## 4.5 Longitudinal Analysis of Change From Baseline

#### **4.5.1** Mixed Model Repeated Measures

Change from baseline in PRO domain (single or multi-item) and overall scores while on study drug treatment will be further analyzed using a restricted maximum likelihood (REML)-based repeated measures approach (MMRM – Mixed Model Repeated Measures) (Brown & Prescott, 2006).

The MMRM assumes that the missing observations are missing at random (MAR). That is, MMRM assumes that, given the statistical model and given the observed values of the outcome, missingness is independent of the unobserved values. A corollary is that MAR assumes that a subject's missing values can be estimated based on similar subjects who remained in the study. This infers that withdrawals (who may not receive study medication) have similar symptoms to some who continue to be treated. While MAR's assumption of the similarity of withdrawals and those who stay in the study may not be realistic for all subjects, MAR can be justified as not being biased to an important degree in favor of the zolbetuximab arm. Given that subjects tend to have poor efficacy scores before they withdraw, MAR will

tend to impute similarly poor symptoms for the missing values: MAR will to that extent reflect that withdrawals are "different" from those who stay in the study.

The primary objective of this analysis is to compare zolbetuximab versus placebo at Cycle 9 Day 1. The Cycle 9 Day 1 timepoint was selected to minimize the impact of missing data given that median rPFS for placebo arm is 12 months (as confirmed by the 8951-CL-0301 study results).

Separate MMRM analysis will be considered for each PRO score:

- QLQ-C30: global health, physical functioning, role functioning, emotional functioning, cognitive functioning, social functioning, fatigue, nausea and vomiting, pain, dyspnea, insomnia, appetite loss, constipation, diarrhea
- QLQ-OG25: Dysphagia, eating restrictions, reflux, odynophagia, pain and discomfort, anxiety, eating in front of others, dry mouth, trouble with taste, body image, trouble swallowing saliva, choked when swallowing, trouble with coughing, trouble talking, weight loss, hair loss
- GP: Pain item
- EQ-5D-5L: EQ-5D-5L utility index (UK mapping algorithm), EQ-5D-5L VAS

The analysis will be based on observed data, i.e., data collected at each time point without carrying forward previous values. Only subjects with a baseline and at least one post-baseline score will be included in the analysis. All visits with at least 10% of patients have non-missing data in each treatment arm will be included, excluding the study discontinuation and safety follow-up visits.

The response variable will be the change from baseline to each post-baseline assessment visit for each PRO score. The model will include the following covariates:

- Fixed effects
  - o Treatment arm (zolbetuximab or placebo)
  - o Timepoint (categorical: visit)
  - o Baseline PRO score (continuous)
  - o Region (Asia vs Non-Asia)
  - o Number of metastatic sites (0 to 2 vs  $\ge$ 3)
  - o Prior gastrectomy (yes vs no)
- Interactions
  - Baseline PRO score x time
  - o Treatment arm x time

Both main effects and the interaction terms will remain in the model, regardless of significance. The model will present least squares (LS) mean estimates, standard errors, 95%

ISN/Protocol 8951-CL-0301

CIs, and p-values (where applicable) for mean changes from baseline to each visit. A plot of the LS means accompanied by the 95% CI will be produced.

In addition, an overall adjusted mean estimate will be derived that will estimate the average change from baseline across all time points, giving each visit equal weight.

The standardized mean difference (SMD) including 95% CI (Hedges' g) will also be provided.

The analysis will be conducted using PROC MIXED in SAS. The model will assume unstructured covariance among the within-subject repeated measurements. If the algorithm does not converge, a heterogeneous Toeplitz (the TOEPH option in SAS PROC MIXED) will be tried first and then AR(1) as a covariance structure to achieve convergence. The Kenward-Roger approximation will be used to estimate denominator degrees of freedom.

Variables listed as categorical in the list above will be included in the CLASS statement of the procedure. The unique subject identifier will also be included as a class variable. A REPEATED statement over the visits will be included with the unique subject identifier as the SUBJECT variable in the REPEATED statement.

The normality and homoscedasticity of the residuals will be visually checked. Particularly, the scatter plot of the residuals versus the predicted endpoint values and the histograms and the normal probability plots of the residuals will be reviewed. Transformation of the raw data will be considered if the graphs of residuals clearly indicate heavily skewed and heteroscedastic distribution of errors.

## 4.6 Responder Analysis

The responder analysis will be performed for all multi-item and single-item scales of the PRO questionnaires. The analysis will be performed on the FAS population and include only participants who have an assessment at baseline and at least one post-baseline assessment. The following descriptive analyses will be performed:

- The proportion of participants with improvement, who were stable, or deteriorated (section 3.2) will be summarized at each post-baseline PRO assessment visit up to including all cycles with at least 10% of patients with a baseline and at least one post-baseline score (excluding the study discontinuation and safety follow-up visits) using both the primary and the sensitivity thresholds. The denominator in this descriptive analysis will be the number of participants with non-missing data at the particular visit.
- A stacked column chart for the distribution of change in response categories from baseline for each scale of both PROs for each post-baseline assessment up to Cycle 9 Day 1 by treatment arms.

## 4.7 Time to Event Analysis

Kaplan-Meier (KM) curves will be used to estimate the distribution of time to deterioration for the PRO total, domain, and item scores for all three definitions described in section 3.3.

The 50th percentile of Kaplan-Meier estimates will be used to estimate the median duration of time to deterioration (in months). A two-sided 95% confidence interval will be provided for these estimates. Median time to deterioration will be compared using stratified log rank test adjusting for randomization stratification factors: region (Asia vs Non-Asia), number of metastatic sites (0 to 2 vs  $\geq$ 3), and prior gastrectomy (yes vs no). A Kaplan-Meier plot by treatment group will be presented.

Additionally, the benefit of zolbetuximab + mFOLFOX6 compared to placebo + mFOLFOX6 will be evaluated by a single hazard ratio (HR) (zolbetuximab vs placebo) with its 95% confidence interval (CI) based on a stratified Cox regression model with Efron's method of tie handling with the same strata as above. The proportional hazards assumption will be tested by examining plots of complementary log( log(survival)) versus log(time). In case departures from the assumption are observed, only the KM and the quartiles of the survival distribution will be presented. For EORTC QLQ-C30 GHS/QoL, PF, and EORTC QLQ-OG25 Pain, time-to-event analysis will be conducted using one-sided tests at the  $\alpha$ =0.025 significance level for consistency with the clinical SAP.

For each of the four instruments (QLQ-C30, QLQ-OG25, GP, and EQ-5D-5L), the HR, p-value, and 95% CI will also be presented graphically on a forest plot.

Kaplan-Meier analysis will be performed using PROC LIFETEST (SAS procedure). Cox proportional hazard regression model will be performed using PROC PHREG (SAS procedure).

Analyses will be performed separately for the following PRO scores:

- QLQ-C30: role functioning, emotional functioning, cognitive functioning, social functioning, fatigue, nausea and vomiting, pain, dyspnea, insomnia, appetite loss, constipation, diarrhea
- QLQ-OG25: Dysphagia, eating restrictions, reflux, odynophagia, anxiety, eating in front of others, dry mouth, trouble with taste, body image, trouble swallowing saliva, choked when swallowing, trouble with coughing, trouble talking, weight loss, hair loss
- GP: Pain item
- EQ-5D-5L: EQ-5D-5L utility index (UK mapping algorithm), EQ-5D-5L VAS.

#### 4.7.1 Sensitivity Analyses

The time to event analyses will be repeated when deterioration is defined using the sensitivity threshold (see section 3.2).

In addition, the analyses using the primary threshold to define deterioration will also be repeated where death (due to any cause) will be counted as an event.

ISN/Protocol 8951-CL-0301

## 4.8 Subgroup Analyses

Analyses on subgroups will be performed for all PRO domains will be performed to determine whether the treatment effect is concordant among subgroups. The following analyses will be performed:

• TTFD, TTCD and TTDD using the primary threshold and excluding death (i.e. 3 definitions).

The analysis will be performed as described in section 4.7. However, to avoid possible issues related to small number of events, subgroup analyses will not be adjusted for the stratification factors used at randomization. Subgroups are defined in section 3.4.

If there are too few events available for a meaningful analysis of a particular subgroup (it is not considered appropriate to present analyses where there are less than 20 events in a subgroup), the HR and 95% CI will not be produced. In this case, only descriptive summaries will be provided.

## 5 SUPPORTING DOCUMENTATION

## 5.1 Appendix A List of Abbreviations

| Abbreviation | Definition |
|--------------|------------------------------------------------------------|
| ANCOVA | Analysis of covariance |
| CLDN | Claudin |
| CI | Confidence interval |
| DCR | Disease control rate |
| DOR | Duration of response |
| ECDF | Empirical cumulative distribution function |
| ECOG | Eastern cooperative oncology group |
| EORTC | European organization for research and treatment of cancer |
| EQ-5D-5L | EuroQoL group-5 dimension-5 level instrument |
| ES | Effect size |
| GEJ | Gastroesophageal Junction |
| GP | Global pain |
| HER2 | Human epidermal growth factor receptor 2 |
| HR | Hazard ratio |
| HRQoL | Health-related quality of life |
| HRU | Health resource utilization (HRU) |
| ICC | Intraclass coefficient |
| ITT | Intent-To-Treat |
| IRC | Independent review committee |
| LS | Least squares |
| MAR | Missing at random |
| MMRM | Mixed Model Repeated Measures |
| ORR | Objective response rate |
| OS | Overall survival |
| PFS | Progression-free survival |
| PGIC | Patient global impression of change |
| PRO | Patient-reported outcome |
| Q1 | First quartile |
| QoL | Quality of life |
| RECIST | Response evaluation criteria in solid tumors |
| REML | Restricted maximum likelihood |
| ROC | Receiver operating characteristic |
| rPFS | Radiographic progression-free survival |
| SAP | Statistical analysis plan |
| SD | Standard deviation |
| SEM | Standard error of measurement |
| SRM | Standardized response mean |
| TTP | Time to progression |
| VAS | Visual analogue scale |

## 5.2 Appendix B QLQ-C30

ENGLISH



#### EORTC QLQ-C30 (version 3)

We are interested in some things about you and your health. Please answer all of the questions yourself by circling the number that best applies to you. There are no "right" or "wrong" answers. The information that you provide will remain strictly confidential.

Please fill in your initials: Your birthdate (Day, Month, Year): Today's date (Day, Month, Year):

| | | Not at | A<br>Little | Quite<br>a Bit | Very |
|---|---|---|---|---|---|
| 1. | Do you have any trouble doing strenuous activities. | | Little | 4.01 | |
| | like carrying a heavy shopping bag or a suitcase? | 1 | 2 | 3 | 4 |
| 2. | Do you have any trouble taking a <u>long</u> walk? | 1 | 2 | 3 | 4 |
| 3. | Do you have any trouble taking a <b>short</b> walk outside of the house? | 1 | 2 | 3 | 4 |
| 4. | Do you need to stay in bed or a chair during the day? | 1 | 2 | 3 | 4 |
| 5. | Do you need help with eating, dressing, washing | | | | |
| | yourself or using the toilet? | 1 | 2 | 3 | 4 |
| Du | uring the past week: | Not at | A | Quite | Very |
| | | All | Little | a Bit | Much |
| 6. | Were you limited in doing either your work or other daily activities? | 1 | 2 | 3 | 4 |
| 7. | Were you limited in pursuing your hobbies or other | | | | |
| | leisure time activities? | 1 | 2 | 3 | 4 |
| 8. | Were you short of breath? | 1 | 2 | 3 | 4 |
| 9. | Have you had pain? | 1 | 2 | 3 | 4 |
| 10. | Did you need to rest? | 1 | 2 | 3 | 4 |
| 11. | Have you had trouble sleeping? | 1 | 2 | 3 | 4 |
| 12. | Have you felt weak? | 1 | 2 | 3 | 4 |
| 13. | Have you lacked appetite? | 1 | 2 | 3 | 4 |
| 14. | Have you felt nauseated? | 1 | 2 | 3 | 4 |
| 15. | Have you vomited? | 1 | 2 | 3 | 4 |
| 16. | Have you been constipated? | 1 | 2 | 3 | 4 |

Please go on to the next page

ENGLISH

| Du | ring the past week: | Not at<br>All | A<br>Little | Quite<br>a Bit | Very<br>Much |
|---|---|---|---|---|---|
| 17. | Have you had diarrhea? | 1 | 2 | 3 | 4 |
| 18. | Were you tired? | 1 | 2 | 3 | 4 |
| 19. | Did pain interfere with your daily activities? | 1 | 2 | 3 | 4 |
| 20. | Have you had difficulty in concentrating on things, like reading a newspaper or watching television? | 1 | 2 | 3 | 4 |
| 21. | Did you feel tense? | 1 | 2 | 3 | 4 |
| 22. | Did you worry? | 1 | 2 | 3 | 4 |
| 23. | Did you feel irritable? | 1 | 2 | 3 | 4 |
| 24. | Did you feel depressed? | 1 | 2 | 3 | 4 |
| 25. | Have you had difficulty remembering things? | 1 | 2 | 3 | 4 |
| 26. | Has your physical condition or medical treatment interfered with your <u>family</u> life? | 1 | 2 | 3 | 4 |
| 27. | Has your physical condition or medical treatment interfered with your <u>social</u> activities? | 1 | 2 | 3 | 4 |
| 28. | Has your physical condition or medical treatment caused you financial difficulties? | 1 | 2 | 3 | 4 |

## For the following questions please circle the number between 1 and 7 that best applies to you $\,$

29. How would you rate your overall health during the past week?

1 2 3 4 5 6 7

Very poor Excellent

30. How would you rate your overall quality of life during the past week?

1 2 3 4 5 6 7

Very poor Excellent

<sup>©</sup> Copyright 1995 EORTC Quality of Life Group. All rights reserved. Version 3.0

**Sponsor: Astellas** ISN/Protocol 8951-CL-0301

Table 8 EORTC QLQ-C30 Scoring Guide (Fayers et al 2001)

| | Abbreviation | Number of items | Item range* | Version 3.0<br>Item<br>numbers |
|---|---|---|---|---|
| Global health status / QoL | | | | |
| Global health status/QoL<br>(revised)† | QL2 | 2 | 6 | 29, 30 |
| Functional scales | | | | |
| Physical functioning (revised)† | PF2 | 5 | 3 | 1 to 5 |
| Role functioning (revised)† | RF2 | 2 | 3 | 6, 7 |
| Emotional functioning | EF | 4 | 3 | 21 to 24 |
| Cognitive functioning | CF | 2 | 3 | 20, 25 |
| Social functioning | SF | 2 | 3 | 26, 27 |
| Symptom scales / items | | | | |
| Fatigue | FA | 3 | 3 | 10, 12, 18 |
| Nausea and vomiting | NV | 2 | 3 | 14, 15 |
| Pain | PA | 2 | 3 | 9, 19 |
| Dyspnoea | DY | 1 | 3 | 8 |
| Insomnia | SL | 1 | 3 | 11 |
| Appetite loss | AP | 1 | 3 | 13 |
| Constipation | CO | 1 | 3 | 16 |
| Diarrhoea | DI | 1 | 3 | 17 |
| Financial difficulties | FI | 1 | 3 | 28 |

<sup>\*</sup> Item range is the difference between the possible maximum and the minimum response to individual items; most items take values from 1 to 4, giving range = 3.

<sup>† (</sup>revised) scales are those that have been changed since version 1.0, and their short names are indicated in this manual by a suffix "2" – for example, PF2.

ISN/Protocol 8951-CL-0301

#### Scoring algorithm

The QLQ-C30 is composed of both multi-item scales and single-item measures. These include five functional scales, three symptom scales, a global health status / QoL scale, and six single items. Each of the multi-item scales includes a different set of items - no item occurs in more than one scale.

The principle for scoring these scales is the same in all cases:

- 1. Estimate the average of the items that contribute to the scale; this is the raw score.
- 2. Use a linear transformation to standardize the raw score, so that scores range from 0 to 100; a higher score represents a higher ("better") level of functioning, or a higher ("worse") level of symptoms.

The technical details are provided below.

If items I1, I2, ... In are included in a scale, the procedure is as follows:

Calculate the raw score (RS) as follows: RS=(I1+I2+ ... +In)/n

Apply the linear transformation as follows:

Functional scales: Scale score =  $(1 - ((RS - 1)/range) \times 100$ 

Symptom scales / items: Scale score =  $(RS - 1)/range \times 100$ 

Global health status/QoL: Scale score =  $(RS - 1)/range \times 100$ 

where range is the difference between the maximum possible value of RS and the minimum possible value. The QLQ-C30 has been designed so that all items in any scale take the same range of values. Therefore, the range of RS equals the range of the item values (see Table 7).

If at least half the components of a scale are present then the scale score will be calculated using the average of all items answered as the raw score; otherwise the score will be set to missing. For single measures, if the item is missing the scale score is set to missing.

An overall summary score has been suggested that can be calculated as (Giesinger et al 2016) the mean of all scales, except for QL2 and FI, i.e.

Physical Functioning + Role Functioning + Social Functioning + Emotional Functioning + Cognitive Functioning + (100-Fatigue) + (100-Pain) + 100-(Nausea and Vomiting) + (100-Dispensea) + (100-Sleeping Disturbances) + (100-Appetite Loss) + (100-Constipation) + (100-Diarrhoea))/13

## 5.3 Appendix C QLQ-OG25



## EORTC QLQ - OG25

Patients sometimes report that they have the following symptoms or problems. Please indicate the extent to which you have experienced these symptoms or problems during the past week. Please answer by circling the number that best applies to you.

| Du | ring the past week: | Not<br>at all | A<br>little | Quite<br>a bit | Very |
|---|---|---|---|---|---|
| 31. | Have you had problems eating solid foods? | 1 | 2 | 3 | 4 |
| 32 | Have you had problems eating liquidised or soft foods? | 1 | 2 | 3 | 4 |
| 33. | Have you had problems drinking liquids? | 1 | 2 | 3 | 4 |
| 14. | Have you had trouble enjoying your meals? | 1 | 2 | 3 | 4 |
| 35. | Have you felt full up too quickly after beginning to eat? | 1 | 2 | 3 | 4 |
| 36. | Has it taken you a long time to complete your meals? | 1 | 2 | 3 | 4 |
| 37. | Have you had difficulty eating? | 1 | 2 | 3 | 4 |
| 38. | Have you had acid indigestion or heartburn? | 1 | 2 | 3 | 4 |
| 19. | Has acid or bile coming into your mouth been a problem? | 1 | 2 | 3 | 4 |
| 40. | Have you had discomfort when eating? | 1 | 2 | 3 | 4 |
| 11. | Have you had pain when you eat? | 1 | 2 | 3 | 4 |
| 12 | Have you had pain in your stomach area? | 1 | 2 | 3 | 4 |
| 43. | Have you had discomfort in your stomach area? | 1 | 2 | 3 | 4 |
| 14. | Have you been thinking about your illness? | 1 | 2 | 3 | 4 |
| 45. | Have you worried about your health in the future? | 1 | 2 | 3 | 4 |
| 46. | Have you had trouble with eating in front of other people? | 1 | 2 | 3 | 4 |
| 47. | Have you had a dry mouth? | 1 | 2 | 3 | 4 |
| 48. | Have you had problems with your sense of taste? | 1 | 2 | 3 | 4 |
| 49. | Have you felt physically less attractive as a result of your disease or treatment? | 1 | 2 | 3 | 4 |

Please go on to the next page

**Sponsor: Astellas** ISN/Protocol 8951-CL-0301

| D | uring the past week: | Not<br>at all | A | Quite<br>a bit | Very<br>much |
|---|---|---|---|---|---|
| 50 | Here you had difficulty swellowing your salive? | 1 | 2 | 3 | 4 |
| 51 | Have you choked when swallowing? | 1 | 2 | 3 | 4 |
| 52 | Have you coughed? | 10 | 2 | 3 | 4 |
| 53 | Have you had difficulty talking? | 1 | 2 | 3 | 4 |
| 54 | Have you worried about your weight being too low? | 1 | 2 | 3 | 4 |
| 55 | Answer this question only if you lost any hair:<br>If so, were you upset by the loss of your hair? | 13 | 2 | 3 | 4 |

#### QLQ-OG25 Scoring algorithm

The QLQ-OG25 is composed of both multi-item domains and single-item measures. Each of the multi-item domains includes a different set of items - no item occurs in more than one domain.

If at least half the components of a domain are present, then the domain score will be calculated using the average of all items answered as the raw score; otherwise the score will be set to missing. For single measures, if the item is missing the domain score is set to missing.

Data are scored as follows according to the algorithm described in the EORTC QLQ-OG25 scoring manual:

#### **Scales:**

Dysphagia: ((Q31+Q32+Q33)/3-1)/3) \* 100

Eating restrictions: ((Q34+Q35+Q36+Q37)/4-1)/3) \* 100

Reflux: ((Q38+Q39)/2-1)/3) \* 100

Odynophagia: ((Q40+Q41)/2-1)/3) \* 100

Pain and discomfort: ((Q42+Q43)/2-1)/3) \* 100

Anxiety: ((Q44+Q45)/2-1)/3) \* 100

#### **Single items:**

Eating in front of others: (Q46-1)/3 \* 100

Dry mouth: (Q47-1)/3 \* 100

Trouble with taste: (Q48-1)/3 \* 100

Body image: ((Q49-1)/3 \* 100

Trouble swallowing saliva: (Q50-1)/3 \* 100 Choked when swallowing: (Q51-1)/3 \* 100 Trouble with coughing: (Q52-1)/3 \* 100

Trouble talking: (Q53-1)/3 \* 100 Weight loss: (Q54-1)/3 \* 100 Hair loss: (Q55-1)/3 \* 100

The algorithms above transform raw scores to a linear scale ranging from 0 to 100, with a high score for scales/single items representing a high level of symptomatology/problems.

ISN/Protocol 8951-CL-0301

## 5.4 Appendix D GP

## III. Global Pain (1 item)



ISN/Protocol 8951-CL-0301

## 5.5 Appendix E EQ-5D-5L

| Under each heading, please tick the ONE box that best describ | es your health TODAY. |
|---|---|
| MOBILITY | |
| I have no problems in walking about | |
| I have slight problems in walking about | |
| I have moderate problems in walking about | |
| I have severe problems in walking about | |
| I am unable to walk about | |
| SELF-CARE | |
| I have no problems washing or dressing myself | |
| I have slight problems washing or dressing myself | |
| I have moderate problems washing or dressing myself | |
| I have severe problems washing or dressing myself | |
| I am unable to wash or dress myself | ā |
| USUAL ACTIVITIES (e.g. work, study, housework, family or leisure activities) | |
| I have no problems doing my usual activities | |
| I have slight problems doing my usual activities | |
| I have moderate problems doing my usual activities | |
| I have severe problems doing my usual activities | |
| I am unable to do my usual activities | |
| PAIN / DISCOMFORT | |
| I have no pain or discomfort | |
| I have slight pain or discomfort | |
| I have moderate pain or discomfort | |
| I have severe pain or discomfort | _ |
| I have extreme pain or discomfort | _ |
| ANXIETY / DEPRESSION | |
| I am not anxious or depressed | |
| I am slightly anxious or depressed | |
| I am moderately anxious or depressed | |
| I am severely anxious or depressed | _ |
| I am extremely anxious or depressed | ā |

2

UK (English) © 2009 EuroQol Group EQ-5D™ is a trade mark of the EuroQol Group

**Sponsor: Astellas** 

ISN/Protocol 8951-CL-0301

. We would like to know how good or bad your health is TODAY.

- · This scale is numbered from 0 to 100.
- 100 means the <u>best</u> health you can imagine.
   0 means the <u>worst</u> health you can imagine.
- . Mark an X on the scale to indicate how your health is TODAY.
- Now, please write the number you marked on the scale in the box below.

YOUR HEALTH TODAY =

3

UK (English) © 2009 EuroQol Group EQ-5D™ is a trade mark of the EuroQol Group

## **6** REFERENCES

| Aaronson et al 1993 | Aaronson N et al (1993). The European Organisation for Research and Treatment of Cancer QLQ-C30: A quality-of-life instrument for use in international clinical trials in oncology. Journal of the National Cancer Institute, pp. 85:365-376. |
|---|---|
| Brown and Prescott 2006 | Brown H and Prescott R (2006). Applied Mixed Models in Medicine. John Wiley and Sons Ltd, 2nd Edition. |
| Cocks et al, 2012 | Cocks, K. & et al, 2012. Evidence-based guidelines for interpreting change scores for the European Organisation for the Research and Treatment of Cancer Quality of Life Questionnaire Core 30. Eur J Cancer, pp. 48:1713-21. |
| Devlin et al, 2017 | Devlin N, Shah K, Feng Y, Mulhern B, van Hout B. Valuing healthrelated quality of Life: An EQ-5D-5L Value Set for England. Health Economics. 2017;1-16. |
| Dolan, 1997 | Dolan P (1997). Modelling valuations for EuroQol health states. Medical Care 35: 1095-1108. |
| Farrar et al, 2000 | Defining the clinically important difference in pain outcome measures. Pain, 2000. 88(3): p. 287-94. |
| Fayers et al, 2021 | Fayers, P., Aaronson, N., Bjordal, K., Groenvold, M., Curran, D., & Bottomley, A. (2001). EORTC QLQ-C30 Scoring Manual (3rd ed.). EORTC. |
| Giesinger et al, 2016 | Giesinger JM et al (2016). Replication and validation of higher order models demonstrated that a summary score for the EORTC QLQ-C30 is robust. J Clin Epidemiol. 2016 Jan;69:79-88. doi: 10.1016/j.jclinepi.2015.08.007 |
| Hernández Alava et al,<br>2017 | Hernández-Alava, M., & Pudney, S. E. (2017). Econometric modelling of multiple self-reports of health states: The switch from EQ-5D-3L to EQ-5D-5L in evaluating drug therapies for rheumatoid arthritis. Journal of Health Economics, 55, 139–152. |
| Hernández Alava et al,<br>2020 | Hernández Alava, M, Pudney, S., Wailoo, A. (2020) Estimating the relationship between EQ-5D-5L and EQ-5D-3L: results from an English Population Study. Policy Research Unit in Economic Evaluation of Health and Care interventions. Universities of Sheffield and York. Report 063. |
| Kendrick and Strout,<br>2005 | The minimum clinically significant difference in patient assigned numeric scores for pain. Am J Emerg Med, 2005. 23(7): p. 828-32. |
| NICE position statement, 2019 | NICE position statement, available at:<br>https://www.nice.org.uk/Media/Default/About/what-we-do/NICE-guidance/NICE-technology-appraisal-guidance/eq5d5l nice position statement.pdf |
| NICE 2022 | National Institute for Health and Care Excellence (2022) NICE health technology evaluations: the manual Process and methods [PMG36], https://www.nice.org.uk/process/pmg36/resources/nice-health-technology-evaluations-the-manual-pdf-72286779244741 |
| Norman et al 2003 | Norman GR, Sloan JA, Wyrwich KW (2003). Interpretation of changes in health-related quality of life: the remarkable universality of half a standard deviation. Med Care 2003; 41(5): 582–592. |
| Pickard et al, 2007 | Pickard AS, Nearry MP and Cella D. (2007). Estimation of minimally important differences in EQ-5D utility and VAS scores in cancer. Health and quality of life outcomes. 5:70. |

**Sponsor: Astellas** ISN/Protocol 8951-CL-0301 PRO SAP Version 2.0

| Sloan et al 2005 | Sloan JA, Cella D, Hays RD (2005). Clinical significance of patient- |
|---|---|
| | reported questionnaire data: another step toward consensus. J Clin |
| | Epidemiol 2005; 58 (12): 1217–1219. |

**Sponsor: Astellas** ISN/Protocol 8951-CL-0301

## **7** SIGNATURE

